CLINICAL TRIAL: NCT05479734
Title: Promoting Resilience and Lowering Risk in Early Childhood: An mHealth Intervention Study
Brief Title: Promoting Resilience and Lowering Risk in Early Childhood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 13549
Record Dates: First submitted 2022-07-08; First posted 2022-07-29 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Child Abuse; Child Neglect; Parenting; Child Development

STUDY DESIGN:
Intervention Model Description: The statistical model is outcome dependent. Some outcomes were measured at pre-intervention, mid-intervention, and post-intervention assessment points allowing for classic crossover study design analyses of intervention arm differences. Other outcomes were only measured at pre-intervention and post-intervention assessment points and allow for classic within-group pre-post change analyses. Feasibility and usability outcomes were effectively measured at post-intervention only and were analyzed with one-sample Wilcoxon signed rank tests to detect moderate or greater levels of feasibility/utility.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No parenting tip, then parenting tips (Experimental): In this crossover arm, participants are assigned to an EMA Only condition for the first two weeks (14 days) of study involvement. During this time, parents receiving daily alerts to complete an ecological momentary assessment (EMA) that asks participants to provide information on recent parent-child interactions, current stressors or challenges, and their child's emotional and behavioral functioning. For the last two weeks of study involvement (days 15 through 28), this group continues to complete the once-daily EMA survey, but they also receive app-delivered parenting tips twice daily. While in this condition phase, a tip notification is delivered to the participant's mobile phone once in the morning and once in the evening. Participants must click on the notification to reveal the parenting tip within the app interface.
  Interventions: Behavioral: mHealth Intervention
- Parenting tips, then no parenting tips (Experimental): In this crossover arm, participants are assigned to the EMA + mHealth intervention (i.e., app-delivered parenting tips twice daily) condition for the first two weeks (14 days) of study involvement. During this time, parents receiving daily alerts to complete an ecological momentary assessment (EMA) that asks participants to provide information on recent parent-child interactions, current stressors or challenges, and their child's emotional and behavioral functioning. During this time, a tip notification is also delivered to the participant's mobile phone once in the morning and once in the evening. Participants must click on the notification to reveal the parenting tip within the app interface. For the last two weeks of study involvement (days 15 through 28), this group continues to complete the once-daily EMA survey, but the parenting tips are no longer delivered.
  Interventions: Behavioral: mHealth Intervention

INTERVENTIONS:
Behavioral: mHealth Intervention — A smartphone app (mHealth app) will deliver daily tailored messages with tips on monitoring and promoting child development and positive parenting tips.

SUMMARY:
An intervention study to provide in-the-moment parenting tips with the goal of increasing healthy parent-child interactions leading to resiliency in high-risk children. Specifically, in a sample of parents participating in HV programs, the investigators will use a smartphone app (mHealth app) to deliver daily tailored messages with tips on monitoring and promoting child development. Daily assessments of parents' emotions, parenting behaviors, and interactions with their children will also be collected via the app. During the 4-week EMA study, parents will receive either 2 weeks of the mHealth intervention + EMA data collection followed by 2 weeks of only EMA data collection or to receive 2 weeks of only EMA data collection followed by 2 weeks of mHealth intervention + EMA data collection.

DETAILED DESCRIPTION:
This is an intervention study to provide in-the-moment parenting tips with the goal of educating parents about monitoring and promoting child development, thereby increasing healthy parent-child interactions leading to resiliency in high-risk children. Specifically, in a sample of parents participating in a HV program, the investigators will use a smartphone app (mHealth app) to deliver twice-daily tailored messages with tips on monitoring and promoting child development. Ecological momentary assessments (EMA) of parents' emotions, parenting behaviors, and interactions with their children will also be collected via the mHealth app. Building off previous work the investigators expect that parents will evidence greater engagement in positive parenting practices on days when they receive the mobile-based parenting tips and strategies relative to on days when they do not receive this content.

The investigators hypothesize that in-the-moment parenting tips delivered around peak times of parent-child interactions (i.e., before work/school, mealtimes, and bedtime) will promote positive parenting practices in a sample of parents at increased risk of adversity exposure. The investigators aim to use EMA methodology to measure both group level differences (i.e., intervention vs. services as usual) and within-person fluctuations in harsh parenting, children's emotional and behavioral functioning, and positive parenting practices. The study will evaluate the following aims and hypotheses:

Aim 1. Conduct a 2-arm, randomized, controlled crossover trial to examine the feasibility and effectiveness of a mobile-based parenting app with parents participating in HV services.

Hypothesis 1a. Parents will report high rates of satisfaction and usability. Hypothesis 1b. Parents will evidence greater engagement in positive parenting practices on days when they receive the mobile-based parenting tips and strategies relative to days when they do not receive this content.

Hypothesis 1c. Groups will evidence increases in positive parenting subscale scores after a month of app engagement.

Aim 2. Utilize EMA data and follow-up assessments to examine the impact of positive parenting practices on the promotion of child development.

Hypothesis 2a. Children will demonstrate less challenging and more positive behavioral functioning on days when their parents receive positive parenting tips.

Hypothesis 2b. Groups will evidence increases in developmental scores after a month of app engagement.

ELIGIBILITY:
Inclusion Criteria:

* Any new or currently enrolled parent in Oklahoma or Tulsa County in MIECHV-funded home visiting programs.

Exclusion Criteria:

* Parents residing outside of Oklahoma or Tulsa Counties will not be recruited (although if they move to another county between baseline and follow-up, they may be eligible to complete the follow-up survey at the discretion of the Principal Investigator).
* Parents who cannot read/speak English or Spanish at an 8th-grade level or higher will not be recruited.
* Parents under age 16 will not be recruited. Parents ages 16-17 meeting other eligibility requirements may be recruited using the assent form with signatures from both of his/her parents.

Ages: 0 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-11-07 (Actual); Primary Completion 2023-06-12 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bard, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- University of Oklahoma Health Science Center- Center on Child Abuse and Neglect, Oklahoma City, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment of clients involved the assistance of up to 3 home visiting agencies in two urban counties in the SW U.S. All agencies were participating in a quality improvement network focused on developmental monitoring and promotion. Agencies that elected to design QI projects that promoted the study parenting app were asked to deliver an initial study pitch to willing and eligible clients. Clients that opted-in were later contacted by the study team for more comprehensive study recruitment.
Groups:
- No Parenting Tip, Then Parenting Tips: This group is asked to complete a daily survey using the mHealth smartphone app (mHealth app) for the first 14 days of participation. The group will then receive twice daily (once in the morning and once in the evening) parenting tips (tailored messages with tips on monitoring and promoting child development) within the app for another 14 days. Participants continue to complete a daily evening survey during the days they receive parenting tips.
- Parenting Tips, Then no Parenting Tips: The group will receive twice daily (once in the morning and once in the evening) parenting tips (tailored messages with tips on monitoring and promoting child development) within the mHealth smartphone app (mHealth app) for the first 14 days. Participants will also complete a daily evening survey during the days they receive parenting tips. Starting on the 15th day, this group is only asked to complete a daily survey (parenting tips are no longer delivered) using the mHealth smartphone app for another 14 days of participation.
Period: Baseline Assessment
Arm/Group | No Parenting Tip, Then Parenting Tips | Parenting Tips, Then no Parenting Tips
Started | 11 | 13
Completed | 11 | 13
Not Completed | 0 | 0
Period: Week 1 App Use (1+ Survey and/or Tips)
Arm/Group | No Parenting Tip, Then Parenting Tips | Parenting Tips, Then no Parenting Tips
Started | 11 | 13
Completed | 10 | 13
Not Completed | 1 | 0
Not completed — No app interactions logged | 1 | 0
Period: Week 2 App Use (1+ Survey and/or Tips)
Arm/Group | No Parenting Tip, Then Parenting Tips | Parenting Tips, Then no Parenting Tips
Started | 11 | 13
Completed | 11 | 13
Not Completed | 0 | 0
Period: Week 3 App Use (1+ Survey and/or Tips)
Arm/Group | No Parenting Tip, Then Parenting Tips | Parenting Tips, Then no Parenting Tips
Started | 11 | 13
Completed | 11 | 10
Not Completed | 0 | 3
Not completed — No app interactions logged | 0 | 3
Period: Week 4 App Use (1+ Survey and/or Tips)
Arm/Group | No Parenting Tip, Then Parenting Tips | Parenting Tips, Then no Parenting Tips
Started | 11 | 13
Completed | 11 | 8
Not Completed | 0 | 5
Not completed — No app interactions logged | 0 | 5
Period: Post-Intervention Assessment
Arm/Group | No Parenting Tip, Then Parenting Tips | Parenting Tips, Then no Parenting Tips
Started | 11 | 13
Completed | 11 | 12
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | No Parenting Tip, Then Parenting Tips | Parenting Tips, Then no Parenting Tips | Total
Number analyzed (Participants) | 11 | 13 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (6.9) | 31.0 (8.2) | 31.7 (7.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 8 | 17
  Not Hispanic or Latino | 2 | 5 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 10 | 11 | 21
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Positive Parenting Practices: EMA Data Positive Parenting Activity Engagement
Description: Participants select the positive parenting activities they engaged in with their child each day during the EMA study (0 is the lowest and represents no engagement in positive parenting practices and a higher number reflects more activities reported). Analyses compared average activity counts during periods with and without app-delivered parenting tips.
Time Frame: Daily EMA Data (28 days)
Population: Three participants did not provide data on this measure during their No Parenting Tips period.
Measure: Least Squares Mean (Standard Error); unit: Daily number of activities
Groups:
- No Parenting Tips: Represents period of time when participants were not receiving the parenting tips through the app.
- Receiving Parenting Tips: Represents period of time when participants were receiving parenting tips through the app.
Arm/Group | No Parenting Tips | Receiving Parenting Tips
Number analyzed (Participants) | 21 | 24
Daily number of activities | 3.75 (0.25) | 2.38 (0.24)
Statistical Analysis 1: Comparison: No Parenting Tips vs Receiving Parenting Tips; Null hypothesis is the number of positive activities engaged in with the child will not differ during the periods with and without app-delivered parenting tips. Mixed effects models were performed regressing mean activity counts on a 'Tips Active' indicator and a measurement-period (1st two weeks vs last two weeks) indicator; Test type: Superiority — Expected Outcomes: greater number of activities while receiving parenting tips; p < 0.01, Mixed Models Analysis — Test performed with significance level of 0.05 (two-sided); The model coefficient t-test uses Satterthwaite's degrees of freedom. An intervention effect difference by sequence is reported when significant

2. Primary Outcome: Parenting Behavior: Alabama Parenting Questionnaire- Positive Parenting Subscale
Description: The Alabama Parenting Questionnaire contains 3 subscales previously used with parents of young children that represent different dimensions of parenting. Each item is rated on a 1 (never) to 5 (always) Likert scale. A higher score on each subscale represents more engagement in that parenting behavior. This analysis focused on the Positive Parenting Subscale (12 items; score range: 12-60).
Time Frame: Change from baseline to post-intervention
Population: As explained under Study Design, some outcomes were only measured at pre- and post-intervention assessment points and, therefore, only allow for classic within-group pre-post change analyses. This restriction applies to this outcome; thus, no test for differences between the experimental arms was conducted.
  Also, 1 participant skipped too many items at baseline, and a subscale calculation was not warranted. 1 participant did not complete the post-intervention assessment (lost to follow-up).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Baseline Assessment: This arm represents the participant-reported outcome before receiving the parenting-app intervention.
- Post-Intervention Assessment: This arm represents the participant-reported outcome after receiving the parenting-app intervention.
Arm/Group | Baseline Assessment | Post-Intervention Assessment
Number analyzed (Participants) | 23 | 23
Units on a scale | 47.6 (1.28) | 47.6 (1.28)
Statistical Analysis 1: Comparison: Baseline Assessment vs Post-Intervention Assessment; Null hypothesis is that the mean positive parenting subscale score would not change from the baseline to the post-intervention assessment. Mixed effects models were performed regressing mean subscale scores on a timeframe (baseline vs post) indicator and a randomization group (early vs late app-delivered parenting tips) indicator. A randomization group difference over time was evaluated. This interaction effect was not included in the final statistical model unless statistically significant; Test type: Superiority; p < 1.00, Mixed Models Analysis — Test was performed with a significance level of 0.05 (two-sided); The model coefficient t-test uses Satterthwaite's degrees of freedom. A randomization group difference over time is reported if significant

3. Primary Outcome: Positive Parenting Practices: EMA Data Time Spent With Child Daily (in Hours)
Description: Mean number of hours spent with the child daily during the periods with and without app-delivered parenting tips.
Time Frame: Daily EMA Data (28 days)
Population: Three participants did not complete EMA assessments during their No Parenting Tips period.
Measure: Least Squares Mean (Standard Error); unit: Daily number of hours
Arm/Group | No Parenting Tips | Receiving Parenting Tips
Number analyzed (Participants) | 21 | 24
Daily number of hours | 2.82 (0.07) | 2.72 (0.07)
Statistical Analysis 1: Comparison: No Parenting Tips vs Receiving Parenting Tips; Null hypothesis is that the number of hours spent with the child will not differ during the periods with and without app-delivered parenting tips. Mixed effects models were performed regressing mean number of hours on a 'Tips Active' indicator and a measurement-period (1st two weeks vs last two weeks) indicator; Test type: Superiority; p < 0.14, Mixed Models Analysis — Test was performed with a significance level of 0.05 (two-sided); [statistical method as in outcome 1, analysis 1]

4. Primary Outcome: Helped me Interact Positively With Child
Description: Participants responded on a scale from Not at all helpful (scored -1) to Extremely helpful (scored 3).
Time Frame: Post-intervention Assessment
Population: As explained under Study Design, feasibility and usability outcomes were only measured at post-intervention and were analyzed with one-sample Wilcoxon signed rank tests to detect moderate or greater levels of feasibility/utility. This restriction applies to this outcome; thus, no test for differences between the experimental arms was conducted.
  Also, 1 participant skipped this item at the post assessment. 1 participant did not complete the post-assessment (lost to follow-up).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Post-Intervention Assessment
Number analyzed (Participants) | 22
Units on a scale | 1.64 (1.18)
Statistical Analysis 1: Comparison: Post-Intervention Assessment; Null hypothesis was that the app was only slightly helpful (scored 0). A Wilcoxon signed rank test was first performed to evaluate potential differences across randomization groups (early vs late app-delivered parenting tips). When the test of a randomization group difference was not significant, the analysis continued with a one-sample Wilcoxon signed rank test; Test type: Other — The model tested the significance of a non-zero location of the data. Effects significantly greater than zero reflect endorsement of app helpfulness; p < 0.01, Wilcoxon (Mann-Whitney) — Test performed with significance level of 0.05 (two-sided)

5. Primary Outcome: Interest in Using the App in the Future
Description: Participants responded on a scale from Not at all interested (scored -1) to Extremely interested (scored 3).
Time Frame: Post-Intervention Assessment
Population: As explained under Study Design, feasibility and usability outcomes were only measured at post-intervention and were analyzed with one-sample Wilcoxon signed rank tests to detect moderate or greater levels of feasibility/utility. This restriction applies to this outcome; thus, no test for differences between the experimental arms was conducted.
  Also, 1 participant skipped this item. 1 participant did not complete the post-assessment (lost to follow-up).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Post-Intervention Assessment
Number analyzed (Participants) | 22
Units on a scale | 1.41 (1.26)
Statistical Analysis 1: Comparison: Post-Intervention Assessment; Null hypothesis was that there would only be slight interest (scored 0) in using the app in the future. A Wilcoxon signed rank test was, first, performed to evaluate potential differences across randomization groups (early vs late app-delivered parenting tips). When the test of a randomization group difference was not significant, the analysis continued with a one-sample Wilcoxon signed rank test; Test type: Other — The model tested the significance of a non-zero location of the data. Effects significantly greater than zero reflect endorsement of future app use; p < 0.01, Wilcoxon (Mann-Whitney) — Test performed with significance level of 0.05 (two-sided)

6. Primary Outcome: Recommend the App to a Friend
Description: Participants responded on a scale from Extremely unlikely (scored -3) to Extremely likely (scored 3).
Time Frame: Post-Intervention Assessment
Population: As explained under Study Design, feasibility and usability outcomes were only measured at post-intervention and were analyzed with one-sample Wilcoxon signed rank tests to detect moderate or greater levels of feasibility/utility. This restriction applies to this outcome; thus, no test for differences between the experimental arms was conducted.
  1 participant did not complete the post-assessment (lost to follow-up).
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Post-Intervention Assessment
Number analyzed (Participants) | 23
Units on a scale | 1.48 (1.81)
Statistical Analysis 1: Comparison: Post-Intervention Assessment; Null hypothesis was that the participant was neither likely nor unlikely (scored 0) to recommend the app to friends. A Wilcoxon signed rank test was, first, performed to evaluate potential differences across randomization groups (early vs late app-delivered parenting tips). When the test of a randomization group difference was not significant, the analysis continued with a one-sample Wilcoxon signed rank test; Test type: Other — The model tested the significance of a non-zero location of the data. Effects significantly greater than zero reflect a desire to recommend the app; p < 0.01, Wilcoxon (Mann-Whitney) — Test performed with significance level of 0.05 (two-sided)

7. Secondary Outcome: General Child Development Score
Description: Developmental Profiles-4 parent/caregiver interview contains five subscales: social-emotional, physical, communication, cognitive, and adaptive behavior. Each subscale score is age standardized with an average of 100 and a standard deviation of 15 (minimum score of 40, maximum score of 160). The General Development Score used in this analysis represents a standardized composite of the 5 subscale scores (minimum score of 46, maximum score of 150). A higher composite score indicates more advanced child development.
Time Frame: Change from baseline to post-intervention
Population: As explained under Study Design, some outcomes were only measured at pre- and post-intervention assessment points and, therefore, only allow for classic within-group pre-post change analyses. This restriction applies to this outcome; thus, no test for differences between the experimental arms was conducted. 1 participant did not complete the post-intervention assessment (lost to follow-up).
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Baseline Assessment | Post-Intervention Assessment
Number analyzed (Participants) | 24 | 23
Units on a scale | 99.6 (3.92) | 101.0 (3.94)
Statistical Analysis 1: Comparison: Baseline Assessment vs Post-Intervention Assessment; Null hypothesis is that the mean general development scale score would not change from the baseline to the post-intervention assessment. Mixed effects models were performed regressing mean scale scores on a timeframe (baseline vs post) indicator and a randomization group (early vs late app-delivered parenting tips) indicator; Test type: Superiority; p < 0.54, Mixed Models Analysis — Test performed with significance level of 0.05 (two-sided); [statistical method as in outcome 2, analysis 1]

8. Secondary Outcome: Child Behavior: EMA Challenging Child Behaviors
Description: Parents report the number of challenging (difficult to manage) child behaviors daily. Analyses compared average behavior counts during periods with and without app-delivered parenting tips.
Time Frame: Daily EMA Data (28 days)
Population: Three participants did not provide EMA data during the No Parenting Tips period.
Measure: Least Squares Mean (Standard Error); unit: Daily number of challenging behaviors
Arm/Group | No Parenting Tips | Receiving Parenting Tips
Number analyzed (Participants) | 21 | 24
Daily number of challenging behaviors | 0.50 (0.06) | 0.33 (0.06)
Statistical Analysis 1: Comparison: No Parenting Tips vs Receiving Parenting Tips; Null hypothesis is that the number of challenging child behaviors will not differ during the periods with and without app-delivered parenting tips. Mixed effects models were performed regressing mean behavior counts on a 'Tips Active' indicator and a measurement-period (1st two weeks vs last two weeks) indicator; Test type: Superiority; p < 0.01, Mixed Models Analysis — Test performed with significance level of 0.05 (two-sided); The model coefficient t-test uses Satterthwaite's degrees of freedom. An intervention effect difference by sequence is reported if significant

9. Secondary Outcome: Child Behavior: EMA Positive Child Behaviors
Description: Parents report the number of positive ("good") child behaviors daily. Analyses compared average behavior counts during periods with and without app-delivered parenting tips.
Time Frame: Daily EMA Data (28 days)
Population: Three participants did not provide EMA data during the No Parenting Tips period.
Measure: Least Squares Mean (Standard Error); unit: Daily number of positive behaviors
Arm/Group | No Parenting Tips | Receiving Parenting Tips
Number analyzed (Participants) | 21 | 24
Daily number of positive behaviors | 2.54 (0.13) | 2.21 (0.13)
Statistical Analysis 1: Comparison: No Parenting Tips vs Receiving Parenting Tips; Null hypothesis is that the daily number of positive child behaviors will not differ during the periods with and without app-delivered parenting tips. Mixed effects models were performed regressing mean behavior counts on a 'Tips Active' indicator and a measurement-period (1st two weeks vs last two weeks) indicator; Test type: Superiority — Expected Outcomes: greater number of behaviors while receiving parenting tips; p < 0.01, Mixed Models Analysis — Test performed with significance level of 0.05 (two-sided); [statistical method as in outcome 8, analysis 1]

ADVERSE EVENTS:
Time Frame: Participants were followed for up to 3 months as they completed a baseline assessment, 1 month of app interaction, and a post-intervention assessment.
Arm/Group | No Parenting Tip, Then Parenting Tips | Parenting Tips, Then no Parenting Tips
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/13
Other Adverse Events (participants affected / at risk) | 0/11 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT05479734/Prot_SAP_000.pdf